CLINICAL TRIAL: NCT00828789
Title: A Phase I, Open-label, Randomized, Crossover Trial in 20 Healthy Subjects to Investigate the Pharmacokinetic Interactions Between the Combination of Efavirenz and Tenofovir Disoproxil Fumarate and Different Dosages of Telaprevir.
Brief Title: VX-950-TiDP24-C134: Drug-drug Interaction Trial Between Combination of Efavirenz and Tenofovir Disoproxil Fumarate and Different Dosages of Telaprevir on Healthy Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR015790
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Hepatitis C; HCV; HIV; AIDS
Keywords: Hepatitis C; HCV; HIV; AIDS; Telaprevir; Efavirenz; Tenofovir disproxil fumarate; Healthy volunteer; VX-950-C134; VX-950-TiDP24-C134; HIV Infections
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — efavirenz; Tenofovir; telaprevir

INTERVENTIONS:
Drug: Efavirenz; Tenofovir disoproxil fumarate; Telaprevir

SUMMARY:
The purpose of this study is to determine the effect of EFV (Efavirenz) and TDF (Tenofovir disoproxil fumarate) on the pharmacokinetics of TVR (Telaprevir) and to determine the effect of TVR on the pharmacokinetics of EFV and TDF. Pharmacokinetics means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body. Furthermore, the short-term safety and tolerability of giving TVR, EFV and TDF together will be evaluated.

DETAILED DESCRIPTION:
The trial will enroll 20 Healthy volunteers. All participants will receive 4 different treatments:

Treatment A: TVR every 8 hours alone for 6 days with an additional morning intake on Day 7. Treatment B: EFV + TDF once daily alone for 7 days. Treatment C: TVR every 8 hours + EFV once daily + TDF once daily for 7 days. Treatment D: TVR every 12 hours + EFV once daily + TDF once daily for 7 days.

All participants will start with Treatment A followed by a 7 or 8-day washout period. Subsequently, participants will start with Treatment B. At the end of Treatment B, participants will be randomized (this is assigned to one of the two sequences by chance) to continue without a washout period with Sequence 1 (Treatment C followed by D without a washout) or Sequence 2 (Treatment D followed by C without a washout). Participants will thus receive daily EFV and TDF for a total of 21 consecutive days, with addition of 2 different dosages of TVR for the last 14 days.

TVR will be taken with food, 30 minutes after the start of a meal. EFV and TDF should be taken on an empty stomach (2.5 hours after start of breakfast). Pharmacokinetic profiles of TVR and VRT-127394 (R-diastereomer of TVR) will be measured up to 8 hours after intake of the morning dose on Day 7 of Treatments A and C, and up to 12 hours after intake of the morning dose on Day 7 of Treatment D. Pharmacokinetic profiles of EFV and tenofovir will be measured up to 24 hours after intake on Day 7 of Treatments B, C, and D. Safety and tolerability evaluations will be recorded at regular intervals throughout the trial period. Treatment A: TVR every 8 hours alone for 6 days with an additional morning intake on Day 7. Treatment B: EFV + TDF once daily alone for 7 days. Treatment C: TVR every 8 hours + EFV once daily + TDF once daily for 7 days. Treatment D: TVR every 12 hours + EFV once daily + TDF once daily for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Females should be post-menopausal (amenorrheal for at least 3 years), or have undergone tubal ligation (or other permanent birth control methods), or hysterectomy (total), or oophorectomy (bilateral)
* Normal weight at screening as defined by a body mass index (BMI, weight in kg divided by the square of height in meters) of 18 to 30 kg/m2, extremes included
* Normal 12-lead ECG at screening
* Healthy on the basis of a physical examination, medical history, ECG, vital signs, and the results of blood biochemistry, blood coagulation and hematology tests and a urinalysis carried out at screening
* Nonsmoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months before study screening.

Exclusion Criteria:

* No history or presence of relevant drug or food allergies, cardiovascular or central nervous system disease, clinically significant pathology, mental disease or psychiatric disorders, chronic skin disease, or drug abuse
* Current use of prescription medication
* Regular treatment with over-the-counter medications
* Consumption of herbal medications or dietary supplements
* A history of drug or alcohol abuse or addiction within 2 years prior to dosing, or a positive test for alcohol or drugs
* Participation in a clinical study within 2 months or 5 half lives of the investigational drug prior to the screening visit
* No positive HIV test or hepatitis A, B or C infection
* Having any history of renal disease
* Male subjects with female partners that are pregnant, or planning to become pregnant during the study or within 90 days of the last dose of study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary objectives are to determine the effect of EFV and TDF on the pharmacokinetics of TVR and VRT-127394 and of TVR every 8h and every 12h on the pharmacokinetics of EFV and TDF.

SECONDARY OUTCOMES:
The secondary objective is to determine the short-term safety and tolerability of the coadministration of TVR, EFV and TDF.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA